CLINICAL TRIAL: NCT06748820
Title: E-CANE: a National Program of Remote Health Education Workshops for Adolescents and Young Adults With Cancer
Brief Title: E-CANE: a National Program of Remote Health Education Workshops
Acronym: E-CANE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24OncoHémato01
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Remote Therapeutic Patient Education (e-TPE): TPE is a set of practices aiming at allowing a patient to acquire and preserve abilities and skills to manage actively their disease, cares, and surveillance, in collaboration with the caregivers
  Interventions: Behavioral: Remote Therapeutic Patient Education (e-TPE)

INTERVENTIONS:
Behavioral: Remote Therapeutic Patient Education (e-TPE) — TPE is a set of practices aiming at allowing a patient to acquire and preserve abilities and skills to manage actively their disease, cares, and surveillance, in collaboration with the caregivers

SUMMARY:
About 2000 adolescents and young adults (AYA) are diagnosed with cancer each year in France. This period of life is marked by a maturation and transition phase in various areas (psychological, physical, sexual, socio-professional...). Cancer occurrence has a very particular impact. AYAs diagnosed and treated for cancer have specific medical and psychosocial needs.In response to these specific needs, Therapeutic Education (TPE), initially developed for patients with chronic disease to help them acquire and maintain skills needed to better manage their daily lives with the constraints of their disease and its treatments, has now its place in cancerology. It has been shown to promote patient independence, improve therapeutic adherence (which is particularly poor in adolescents with cancer), and strengthen the therapeutic alliance between patients and their healthcare team. The strengthening of adolescents's self-care and adaptation skills is also recognized as essential during the experience of an oncological disease. In addition, over the past few years, in the context of the increasing use of the internet and digital technologies, particularly in the daily lives of young people, the implementation of remote TPE sessions (e-TPEs) has developed significantly. In cancerology, digital health interventions have the potential to expand access to the support available to youth with cancer. E-health offers flexibility to the delivery of psychosocial care and could help strengthen youth engagement and enable them to interact with professionals and other young people in a reassuring digital context.This project aims to demonstrate the feasibility of conducting remote health education workshops (e-TPE) for AYAs with cancer, regardless of their place of care in French territory. Following an educational assessment conducted by a professional trained in TPE, three digitalized workshops from the DYNAMO program, will be offered. The adherence to this type of educational interventions, the satisfaction of the patients and the professionals involved, but also the obstacles and difficulties encountered will be analyzed. Demonstrating the feasibility of these e-workshops would allow the spread and the enrichment of this type of interventions. This could facilitate their accessibility for all AYAs in French territory. At the end of this experiment, a randomized study could provide scientific evidence that the development of such a program is a relevant strategy to help young people with cancer manage the challenges associated with their diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cancer diagnosed for at least one month.
* Patient followed by an AYA Coordinating Nurse in one of the 27 French AYA centres.
* Patient with Life expectancy ≥ 6 months.
* Patient ealth status consistent with program requirements.
* Karnosky index > 60%.
* Patient who agrees to participate in the program and benefits from social security.
* Patient able to understand, speak and read French.
* Patient with no major cognitive impairment (assessed by the patient's referees).
* Patient with no sensory disability.
* Patient with access to a computer tool (smartphone, tablet, computer) and a WiFi or 4G network.
* Non opposition from patient or their legal representative collected.
* Patient who has signed the Privacy Policy.
* Patient who consented to participate in PTE program.

Exclusion Criteria:

* Patient unable to use informatic tools.
* Known superior cognitive function disorders.
* Progressive psychiatric pathology
* Drug user or alcohol abuse

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and young adults between 15 and 25 years old with cancer followed in a French AYA center.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the patient's adherence to the implementation of remote health educational actions (e-TPE), in AYA patients with cancer undergoing treatment | Between 2 and 4 times over 18 months
  Online self-administered satisfaction questionnaires filled out by the patients 70 questions, scores between 1 and 4, yes or no, multiple choice questions, open-ended questions.

SECONDARY OUTCOMES:
Assess the suitability of the pedagogical methods | 3 times over 12 months
  Online self-administered satisfaction questionnaires filled out by the workshop hosts (12 questions) No scores, yes or no, open-ended questions.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France